CLINICAL TRIAL: NCT05213273
Title: TUNACAN: Nutritional Study on the Beneficial Effects of Canned Fish Consumption on Healthy Adult Population
Brief Title: Nutritional Study on the Beneficial Effects of Canned Fish Consumption on Healthy Adult Population
Acronym: TUNACAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sara Arranz Martinez (Other)
Collaborators: MUTUALIA S.L. (Unknown); OSARTEN KOOPERATIBA ELKARTEA (Unknown)
Responsible Party: Sponsor-Investigator, Sara Arranz Martinez, Senior Researcher, Fundacion Azti
Organization: Fundacion Azti (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SA-TUN-2021-01
Record Dates: First submitted 2021-11-12; First posted 2022-01-28 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Healthy Diet
Keywords: canned fish; red blood cell membrane lipidomics; omega-3 fatty acids

STUDY DESIGN:
Intervention Model Description: Randomized nutritional intervention clinical trial of 2 parallel groups, in which 150 healthy adults between 18 and 65 years will be recruited.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Fresh/frozen fish (Experimental): Healthy diet based on mediterranean guidelines with specific recommendation of fish intake (3-4 servings/week of fresh or frozen fish or shellfish), excluding the consumption of canned fish.
  Interventions: Behavioral: nutritional guidelines to promote healthy diet and increase fish intake
- Group B: Canned fish (Experimental): Healthy diet based on mediterranean guidelines with specific recommendation of fish intake (3-4 servings/week of fresh or frozen fish or shellfish where at least 1-2 servings will be in the form of canned fish). A selection of canned fish (tuna, sardine, salmon and mackerel) will be administered to each volunteer for the duration of the study.
  Interventions: Behavioral: nutritional guidelines to promote healthy diet and increase fish intake

INTERVENTIONS:
Behavioral: nutritional guidelines to promote healthy diet and increase fish intake — Nutritional guidelines based on the Mediterranean diet will be provided to both groups (gropu A and group B) through infographic material, recipes and menus.
  Both groups will be guided to increase their fish consumption to 3 servings per week. Group A will do that through the consumption of fresh or frozen fish and group B through fresh, frozen and canned fish.

SUMMARY:
There is sufficient evidence on the beneficial effects of fish consumption on health, mainly associated with the content of omega-3 polyunsaturated fatty acids (EPA and DHA) present mainly in blue fish. Different national and international organizations have issued recommendations on the optimal amount of fish that the population should consume to prevent certain chronic diseases related to diet. Thus, the WHO recommends eating fish regularly (1-2 servings per week for healthy adults) to ideally provide the equivalent of 250 mg of omega-3 fatty acids (EPA + DHA). Not reaching the optimal levels of EPA + DHA increases the risk for cardiovascular diseases, increasing the risk of death according to certain epidemiological studies. In this sense, using more precise techniques such as membrane lipidomics, allow adequate quantification and monitoring of fatty acid levels present in our body and how this lipid profile can change according to metabolism and diet. The objective of this study is to carry out a clinical trial of nutritional intervention with an adult population without pathologies that has a low consumption of fish (<2 servings / week) to evaluate the effectiveness of an intervention strategy based on increasing the number of fish servings through a controlled intake of fresh and canned fish.

The results aim to show that increasing fish intake has an impact on lipid metabolism and in the future, for the prevention of certain chronic diseases, the introduction of canned fish can be a healthy strategy to increase fish consumption to long term.

DETAILED DESCRIPTION:
Objectives:

The main objective of this study is to demonstrate through a nutritional intervention, the benefits of the intake of canned fish compared to fresh or frozen fish on lipid metabolism in a healthy adult population, which can be divided into three specific objectives:

* Assessment of the health benefits of consuming canned fish (controlled intake): impact on the fatty acid profile of red blood cell membrane.
* Provide evidence of the benefits of consuming canned fish compared to intake fresh / frozen fish.
* Demystify the bad reputation of canned fish products (as processed foods).

Study design:

A prospective, randomized, controlled, parallel-group nutritional intervention clinical trial will be carried out with 150 healthy adults between 18 and 65 years for 4 months. Participants will be randomized into one of the two equal size intervention groups: "group A: fresh/frozed fish" or "group B: canned fish".

Recruitment and selection of participants:

AZTI will organize the selection and recruitment process in collaboration with IMQ-Prevention (MUTUALIA) through 4 centers in Spain (Zamudio, Bilbao, Vitoria and Donosti) and with the OSARTEN Koop clinical analysis laboratory.

Participants will be distributed according to a random assignment sequence. In this way, investigators increase the probability that the two groups (control and intervention) are comparable with respect to age and gender.

Inclusion criteria: Healthy adults (men and women) with 18.5 <BMI < 27 kg/m2. Those individuals who usually have a fish intake of less than 1-2 servings per week will be included.

Exclusion criteria: Having been diagnosed with concomitant diseases or chronic disease that can modify the results. Having undergone a transplant. Be taking medication and consuming or have consumed omega 3 supplements, vitamins, prebiotics.. in the last 4 months before starting the study. Allergy to fish or any food.

Sample size calculation:

The sample size was calculated with the G * power software based on the defined primary objective of observing differences in the lipid profile of the red blood cell membrane obtained after the ANCOVA test for fixed effects and interactions. A priori investigators expect a mean effect (f = 0.25) for a statistical power of 80.0% (1-β = 0.80) and taking into account that the significance level is 5.0%, it will be necessary to include 64 experimental units in the control group and 64 units in the experimental group that sum 128 experimental units in the study. Taking into account that the expected dropout percentage is around 20.0%, a total of 150 experimental units would be necessary in the study.

Primary outcome:

1. Metabolic status will be evaluated measuring 12 fatty acids in red blood cell membrane (relative %). Omega 3 index (EPA+DHA) as a biomarker of cardiovascular risk and omega-6 omega-3 ratio as biomarker of inflammatory status will be the main outcomes. Investigators will take into accounts the optimal ranges of this fatty acids in red blood cell membranes previously reported in the litearature (Ferreri C et al. 2012. Expert Rev. Mol. Diagn. 12(7), 767-780).

   Secondary outcomes:
2. Biochemical parameters: total cholesterol (mg/dL), HDL cholesterol (mg/dL), LDL cholesterol (mg/dL), triglycerides (mg/dL), glucose (mg/dL), uric acid (mg/dL), creatinine (mg/dL) and liver enzyme activities (GGT, GPT, GOT).
3. Body mass index (kg/m2).
4. Nutrients intake (g/day) from Food Frequency Questionnaire.
5. Physical activity (MET-minutes per week) from International Physical Activity Questionnaire (IPAQ).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (men and women)
* 18.5 <BMI <24.9.
* Individuals who habitually have a lower fish intake1-2 servings/week

Exclusion Criteria:

* Diagnosed with concomitant diseases or chronic disease.
* Have been subjected to transplant.
* Be taking medication
* Consuming or having consumed omega-3 supplements, vitamins, minerals, prebiotics or probiotics 3 months before starting the study. Food allergies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Metabolic status: RBC membrane fatty acid profile. | 4 months
  Twelve fatty acids will by analyzed as representative cluster of the main building blocks of the red blood cell (RBC) membrane glycerophospholipids (palmitic acid, stearic acid, palmitoleic acid, oleic acid, cis-vaccenic acid, eicosapentaenoic acid, docosahexaenoic acid, linoleic acid, dihomo-gamma-linolenic acid (DGLA), arachidonic acid (AA) and two geometrical trans fatty acids (trans elaidic acid and mono-trans arachidonic acid isomer).
  The amount of each fatty acid will be calculated as a percentage of the total fatty acid content in the red blood cell membrane (relative %).
  Omega 3 index (EPA+DHA) as a biomarker of cardiovascular risk and omega-6/omega-3 ratio as biomarker of inflammatory status will be the main outcomes. Investigators will take into accounts the optimal ranges of each of the 12 fatty acids in red blood cell membranes previously reported in the literature (Ferreri C et al. 2012. Expert Rev. Mol. Diagn. 12(7), 767-780).

SECONDARY OUTCOMES:
Biochemical parameters in plasma | 4 months
  Blood cholesterol (mg/dL): total cholesterol, HDL-c and LDL-c Triglycerides (mg/dL) Glucose (mg/dL)

OTHER OUTCOMES:
Nutrients intake (g/day) | 4 months
  Participants in the study will complete a food frequency questionnaire based on the PREDIMED validated questionnaire for the Spanish population (Fernández-Ballart et al, 2010). These questionnaire will be completed at the beginning and after 4 months of intervention to measure change in dietary intake (food groups and nutrients). Information about different food items collected from this questionnaire will be analyzed using DIAL® software to translate their intake into their corresponding energy (kilocalories) and nutrient intake (g/day).
Physical activity (MET-min per week) | 4 months
  Participants in the study will complete the international physical activity questionnaire (IPAQ). IPAQ will be scored using the continuous variable MET minutes a week that represent the amount of energy expended carrying out physical activity. Participants will complete this IPAQ at the beginning and after 4 months of intervention to compare physical activity.
Anthropometric parameters (weight and height) | 4 months
  Weight (kg) and height (m) will be combined to report body mass index (BMI) in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Sara Arranz, PhD, Principal Investigator — Fundacion Azti
Locations (1):
- AZTI, Derio, Bizkaia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sara Arranz ORCID — https://orcid.org/0000-0003-2397-5145
- See also: AZTI web page — https://www.azti.es/en/